CLINICAL TRIAL: NCT02588963
Title: Prevention of Respiratory Infections Among Children Under 3 Years of Age Attending
Brief Title: Prevention of Respiratory Infections Among Children Under 3 Years of Age Attending Daycare Centres
Acronym: PRICAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Principal Investigator, Ana Silva Alexandrino, MSc, Polytechnic Institute of Porto
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PIPorto
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Tract Infections
Keywords: upper respiratory tract infections; lower respiratory tract infections; health promotion; respiratory physiotherapy; infant
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Experimental Group 1 (Experimental): Children whose caregivers were subjected to a health education session
  Interventions: Other: Health education session
- Experimental Group 2 (Experimental): Children who were subjected to nasal clearance protocol
  Interventions: Other: Nasal clearance Protocol
- Experimental Group 3 (Experimental): Children whose caregivers were subjected to health education session and who were subjected to respiratory physiotherapy protocol
  Interventions: Other: Health education session; Other: Nasal clearance Protocol
- Control Group (Placebo Comparator): Children who were not subjected to respiratory physiotherapy protocol for nasal clearance and whose parents were not subjected to health education session
  Interventions: Other: Control

INTERVENTIONS:
Other: Health education session — It was created an education health session regarding the prevention of respiratory infections of children, according to caregivers needs. This session have a theoretical component, addressing especially modifiable risk factors of respiratory infections in children, and a practical component where caregivers can learn and practice nasal clearance techniques, demonstrated by the physiotherapist.
  Arms: Experimental Group 1; Experimental Group 3
Other: Nasal clearance Protocol — Nasal clearance protocol consists on the application of physiological serum in the nostrils of the child, followed by the stimulation of nasal inspiration in order to remove mucus from the nose and nasopharynx. The protocol is applied for 3 consecutive days, according to established criteria suggested by Postiaux.
  Arms: Experimental Group 2; Experimental Group 3
Other: Control — Children proceeded to their normal activities at the daycare; Caregivers did not attend to education health session.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the influence of Primary and Secondary Prevention of Respiratory Infections in children up to 3 years-old attending daycare.

DETAILED DESCRIPTION:
Randomized controlled clinical trial including children up-to 3 years-old who attend daycare centres in O Porto.

To evaluate the Primary Prevention of Respiratory infections it was created and ministered to children's caregivers an education health session, regarding the prevention of respiratory infections of children, according to caregivers needs.

It is known that parental perceptions influence their behaviour in respect to the care of their unwell child. Sometimes misunderstandings occurred because parents' expressions of concern or requests for additional information were sometimes perceived as a challenge to the clinicians' diagnosis or treatment decision, which leads to unnecessary and unwanted prescribing of antibiotics. Health professionals should provide consistent information that promotes parental self-efficacy in the care of their unwell child.

To evaluate the Secondary Prevention of Respiratory Infections it was applied to children with signs of upper respiratory infections (rhinorrhea, cough and nasal obstruction) a nasal clearance protocol, developed by Guy Postiaux. This protocol consists on the application of physiological serum in the nostrils of the child, followed by forced nasal inspiration. The protocol is applied for 3 consecutive days, according to established criteria suggested by Postiaux. This intervention is indicated on Upper Respiratory Infections, such as rhinitis or rhinopharyngitis, with large amount of secretions in the upper airway and it is an effective adjuvant for medication. Forced nasal inspiration is able to create sufficient gas velocity to act on the pressure of the middle ear, through the eustachian tube, and may have an important role in the prevention of otitis.

ELIGIBILITY:
Inclusion Criteria: Children of both genders up to 3 years, born at term, pregnancy without complications, attending day care, residents in OPorto, with medical approval for intervention

Exclusion Criteria: Children born prematurely, with lower respiratory infections, with chronic neurological, musculoskeletal, cardiac or respiratory disorders

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Health Indicators | 1 month after intervention
  health status of the child was reported by caregivers concerning the number of episodes of respiratory infections and/or otitis.

SECONDARY OUTCOMES:
Severity of respiratory infection | 1 month
  Paediatric Respiratory Severity Score (PRSS) adapted for the Portuguese culture (Cronbach's alpha = 0.80 and ICC 2,1 = 0.91) was used to assess the child's respiratory clinical parameters, such as dyspnea, breathing sounds, adventitious sounds, daily expectoration, cough, nutrition, fever and rhinorrhea.
Middle Ear Condition | 1 month
  Pressure, compliance and tympanogram of the middle ear were assessed by tympanometry, performed by an audiologist (Hand Held Impedance Audiometer MT10 (Interacoustics1 USA) calibrated on November 22, 2010, according to Food and Drug Administration (FDA) requirements, with a 226 Hz probe tone)
Nasal Auscultation | 1 month
  Pressure, compliance and tympanogram of the middle ear were assessed by tympanometry, performed by an audiologist (Hand Held Impedance Audiometer MT10 (Interacoustics1 USA) calibrated on November 22, 2010, according to Food and Drug Administration (FDA) requirements, with a 226 Hz probe tone)

OTHER OUTCOMES:
Caregivers' Anxiety | 2 months
  Portuguese Version of the Self-rating Zung's Anxiety Scale (r=0,782; ICC=0,95) was applied to caregivers
Caregivers' Knowledge about Respiratory Infections | 2 months
  Written evaluation form was applied to caregivers in order to assess their knowledge about respiratory infections, designed by an expert panel.
Health resources | 1 month
  frequency of use of health resources and/or medication
Absenteeism | 1 month
  number of days that the child were absent at the daycare and/or caregivers were absent at work;

CONTACTS AND LOCATIONS:
Overall Officials: Ana S Alexandrino, MSc, Principal Investigator — School of Allied Health Technologies of the Polytechnic Institute of Porto
Locations (1):
- School of Allied Health Technologies of the Polytechnic Institute of Porto, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ingram J, Cabral C, Hay AD, Lucas PJ, Horwood J; TARGET team. Parents' information needs, self-efficacy and influences on consulting for childhood respiratory tract infections: a qualitative study. BMC Fam Pract. 2013 Jul 28;14:106. doi: 10.1186/1471-2296-14-106. PMID 23890343
- [Background] Cabral C, Horwood J, Hay AD, Lucas PJ. How communication affects prescription decisions in consultations for acute illness in children: a systematic review and meta-ethnography. BMC Fam Pract. 2014 Apr 8;15:63. doi: 10.1186/1471-2296-15-63. PMID 24708839
- [Background] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404
- [Background] Postiaux G, Souza Pinto V, Vieira DR, Carvalho CM. Fisioterapia respiratória pediátrica: o tratamento guiado por ausculta pulmonar. Porto Alegre: Artmed Editora; 2004.
- [Background] Tome D, Alexandrino AM, Santos RI, de Melo MC, Costa DA, Ferreira JP. Characterization of middle-ear condition of Oporto daycare children up-to 3 years-old: a cross sectional study. Int J Pediatr Otorhinolaryngol. 2014 Dec;78(12):2132-5. doi: 10.1016/j.ijporl.2014.09.022. Epub 2014 Sep 30. PMID 25441605
- [Background] Santos R, Silva Alexandrino A, Tome D, Melo C, Mesquita Montes A, Costa D, Pinto Ferreira J. Inter- and intra-rater reliability of nasal auscultation in daycare children. Minerva Pediatr. 2018 Feb;70(1):20-26. doi: 10.23736/S0026-4946.17.04355-9. Epub 2015 Sep 11. PMID 26365822
- [Derived] Alexandrino AS, Santos R, Melo C, Bastos JM. Impact of caregivers' education regarding respiratory infections on the health status of day-care children: a randomized trial. Fam Pract. 2016 Oct;33(5):476-81. doi: 10.1093/fampra/cmw029. Epub 2016 Apr 30. PMID 27131288